CLINICAL TRIAL: NCT03948893
Title: Neural Mechanisms Mediating Appetitive Regulation and Smoking in Nicotine Addiction
Brief Title: Smoking Cessation Behavioral Treatment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Brett Froeliger, Professor Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020602
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MORE (Experimental)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE)
- CBT (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE) — MORE is a behavioral therapy that integrates mindfulness training to modify reward processes.
  Arms: MORE
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT is a therapy designed to help individuals understand how their thoughts and feelings influence their behaviors.
  Arms: CBT

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two behavioral interventions on smoking behavior - Mindfulness-Oriented Recovery Enhancement (MORE) and Cognitive Behavioral Therapy (CBT). MORE is a behavioral therapy that integrates mindfulness training to modify reward processes. CBT is a therapy designed to help individuals understand how their thoughts and feelings influence their behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up
* English fluency as demonstrated in providing informed consent and the ability to independently follow directions in completing assigned assessments and tasks
* Functional vision (with corrective lenses as needed) to complete assigned assessments and tasks
* Current nicotine dependent smoker with a minimum smoking history of 2 years
* Interest in quitting smoking

Exclusion Criteria:

* Use of psychotropic (e.g. antiepileptic) medications in the past month
* Positive urine drug screen
* Presence of an untreated medical illness
* Current or past psychosis
* History of major neurological illness or head injury resulting in loss of consciousness
* And contraindication to MRI, including claustrophobia
* Among females, positive urine pregnancy test
* Inability or unwillingness of subject to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Smoking | 7 weeks
  Biochemical smoking assessment (breath carbon monoxide) at each study visit.
Magnitude of change in fMRI brain response to images | 7 weeks
  Measure the effects of MORE on fMRI BOLD response to images (change from baseline to end of study) while participants undergo functional magnetic resonance imaging
Magnitude of change in fMRI brain connectivity | 7 weeks
  Measure the effects of MORE on resting-state functional connectivity (change from baseline to end of study) while participants undergo functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Missouri - Columbia, Columbia, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No